CLINICAL TRIAL: NCT01998568
Title: The Variation of the Intraocular Pressure Measured by Different Tonometers in Patients With Clinical Corneal Edema
Brief Title: The Intraocular Pressure Measured by Different Tonometers in Corneal Edema
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Doctor, Prince of Songkla University
Other Study IDs: 56-451-02-1
Record Dates: First submitted 2013-11-23; First posted 2013-12-02 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Intraocular Pressure; Corneal Edema
Keywords: Intraocular pressure; Corneal edema; Tonometer; Dynamic contour tonometer; Tonopen; iCare; Goldmann applanation
MeSH Terms: conditions — Corneal Edema | interventions — Intraocular Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Corneal edema: Intraocular pressure measurement
  Interventions: Other: Intraocular pressure measurement

INTERVENTIONS:
Other: Intraocular pressure measurement — Using different tonometers for intraocular pressure measurement

SUMMARY:
The investigators conduct this study to access the effect of corneal edema (the investigators are particularly interested in those who have the clinical central corneal edema) on the variation of intraocular pressure values measured by 3 commercial-available tonometers compare to the current gold standard tonometer; Goldmann applanation tonometer.

DETAILED DESCRIPTION:
Previous published articles reported on the effect of corneal edema on the accuracy of tonometry were performed in enucleated cadaver eyes, or contact lens-induced corneal edema eyes. Thus, it remains unclear as to how the clinical corneal edema that is found in routine clinical practice will affect the variation of intraocular pressure measurement using the standard Goldmann applanation tonometer and other more modern tonometers such as the dynamic contour tonometer, the iCare, and the Tonopen.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 year-old
* Patients who have a clinical central corneal edema after clear cornea phacoemulsification and intraocular lens implantation
* Agree to participate in the study and willing to sign an informed consent

Exclusion Criteria:

* Combined phacoemulsification and trabeculectomy
* Clear cornea phacoemulsification that has suture on the cornea
* Previous history of intraocular surgery, ocular trauma prior to phacoemulsification
* Vitrectomized eye
* History of glaucoma or ocular hypertension or using IOP lowering medication
* History of diabetic retinopathy staged as severe non-proliferative or worse
* Pregnant or breast-feeding women
* History of refractive surgery or any keratoplastic procedure
* Corneal opacities or diseases making no suitable tonometry
* Severe dry eye syndrome
* Wears contact lenses
* Astigmatism higher than 2.5 diopters
* Microphthalmos or buphthalmos
* Subjects with having poor or eccentric fixation or nystagmus
* Excessive eye squeezing
* Known allergy to topical anesthesia
* Known allergy to fluorescein solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a clinical central corneal edema after clear cornea phacoemulsification and intraocular lens implantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | A day after cataract surgery and when the corneal edema is resolve (usually within 1-2 weeks post operatively)
  The intraocular pressure measured by each tonometer compare with Goldmann applanation tonometer (When measure in eyes with corneal edema and when the edema is clinically resolve)

SECONDARY OUTCOMES:
Relationship between the central corneal thickness and intraocular pressure measured by each tonometer | A day after surgery (clinical corneal edema was detected) and within 1-2 weeks (resolution of edema)
  The severity of corneal edema may affect the reliability of intraocular pressure measurement measured by different tonometers

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No